CLINICAL TRIAL: NCT06088901
Title: Utilization of Prophylactic Autologous Blood Patch Pleurodesis in the Treatment of Primary Spontaneous Pneumothorax
Brief Title: Autologous Blood Patch for Primary Spontaneous Pneumothorax
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to screen d/t schedule
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brian Gulack, Assistant Professor, Rush University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23030702
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Primary Spontaneous Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Intervention Model Description: All patients presenting with first occurrence of a PSP who meet criteria for chest tube placement, between the ages of 13-18, will be offered inclusion in Arm 1.
  All patients presenting with recurrent PSP who meet criteria for blebectomy with a pleural procedure, between the ages of 13-18, will be offered inclusion in Arm 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: First Occurrence (Experimental): All patients who meet criteria and consent to involvement will be treated per institutional protocols with a tube thoracostomy. Chest tube size will be determined by the physician of record. Once the chest tube is placed, it will be placed to suction for a minimum of two minutes to allow for lung re-expansion while 2 ml/kg of whole blood (max 100 ml) is obtained via venipuncture (preferably a previously established intravenous catheter). This blood will then be injected via the chest tube which will then be clamped for 180 minutes, before being returned to suction. During this period of clamping, the patient will be rotated from side to side intermittently to help the blood move around the extrapleural space.
  Interventions: Procedure: Autologous Blood Patch
- Arm 2: Recurrence (Experimental): All patients who meet criteria and provide informed consent will be treated per institutional protocols with a thoracoscopic blebectomy and mechanical pleurodesis or pleurectomy. At the conclusion of the procedure, 2 ml/kg of whole blood (max 100 ml) obtained via venipuncture will be injected into the pleural space. The chest tube will be left clamped for 180 minutes post-procedure and then placed back to suction. During this period of clamping, the patient will be rotated from side to side intermittently to help the blood move around the extrapleural space.
  Interventions: Procedure: Autologous Blood Patch

INTERVENTIONS:
Procedure: Autologous Blood Patch — 2 ml/kg of whole blood (max 100 ml) is obtained via venipuncture. This blood is then injected via the chest tube which will then be clamped for 180 minutes, before being returned to suction. During this period of clamping, the patient will be rotated from side to side intermittently to help the blood move around the extrapleural space.

SUMMARY:
The purpose of this study is to show that treatment with prophylactic autologous blood patch (ABP) after management of primary spontaneous pneumothorax (PSP) is feasible, reduces the incidence of prolonged air leaks, and reduces hospital length of stay. An ABP is a medical procedure that uses one's own blood in order to close one or many holes identified in the lungs. The blood modulates the pressure of the lungs and forms a clot, sealing the leak. Primary spontaneous pneumothorax is an abnormal collection of air in the pleural space between the lung and the chest wall.

DETAILED DESCRIPTION:
The investigators will employ a novel treatment algorithm using a previously described technique to determine its feasibility and efficacy. This study will provide necessary quantitative and qualitative data to plan and obtain additional investigator-initiated funding to perform future comparative studies.

ARM 1 Purpose and Goals: Management of PSP at the initial presentation traditionally involves pleural drainage (although some opt for observation in mild cases). Unfortunately, prolonged pulmonary air leaks and recurrence are common, making PSP more consistent with a chronic disease than an acute process. While ABP has traditionally been used in instances of prolonged air leaks after chest tube placement, there is data from other patient populations that routine use at the time of the index procedure may reduce the incidence of prolonged air leaks and consequently patient morbidity and associated costs. The investigators' goal is to demonstrate the feasibility and efficacy of this technique.

Procedures: All patients who meet criteria and consent to involvement will be treated per institutional protocols with a tube thoracostomy. Chest tube size will be determined by the physician of record. Once the chest tube is placed, it will be placed to suction for a minimum of two minutes to allow for lung re-expansion while 2 ml/kg of whole blood (max 100 ml) is obtained via venipuncture (preferably a previously established intravenous catheter). This blood will then be injected via the chest tube which will then be clamped for 180 minutes, before being returned to suction. During this period of clamping, the patient will be rotated from side to side intermittently to help the blood move around the extrapleural space. The remainder of the management will be left to the discretion of the primary physician. The PSP procedure is considered standard of care.

ARM 2 Purpose and Goals: In adolescents who present with recurrent PSP, a resection of the most likely offending bleb as well as a pleural procedure to prevent recurrence is often indicated. Following surgical treatment, patients are hospitalized with a chest tube to manage any persistent air leaks. While the use of an ABP has most commonly been relegated to patients who have persistent air leaks beyond 5 days, previous data has demonstrated benefits of prophylactic ABPs in other pulmonary procedures. The investigators hypothesize that this benefit extends to the surgical management of PSP. The investigators' goal is to demonstrate the feasibility and efficacy of this technique when used prophylactically, in order to provide data for designing a multicenter prospective clinical trial.

Procedures: All patients who meet criteria and provide informed consent will be treated per institutional protocols with a thoracoscopic blebectomy and mechanical pleurodesis or pleurectomy. At the conclusion of the procedure, 2 ml/kg of whole blood (max 100 ml) obtained via venipuncture will be injected into the pleural space. The chest tube will be left clamped for 180 minutes post-procedure and then placed back to suction. During this period of clamping, the patient will be rotated from side to side intermittently to help the blood move around the extrapleural space. The remainder of the post-operative management will be left to the discretion of the primary physician. The PSP procedure is considered standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary spontaneous pneumothorax (first occurrence) and meets criteria for chest tube placement or Diagnosed with recurrent primary spontaneous pneumothorax (recurrence) and meets criteria for blebectomy with a pleural procedure
* Between the ages of 13-18

Exclusion Criteria:

Known hematologic disorders Hemodynamic instability at the time of presentation

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Hospital Length of Stay | 30 days
  Total hospital length of stay will allow a comprehensive evaluation of the efficacy of the intervention. As a continuous variable, this will give the investigators the most power to compare to historical controls. This will take into account not only changes in postoperative air leak but also additional effects from the research intervention.

SECONDARY OUTCOMES:
Incidence of Prolonged Air Leak (>48 hours) | 30 days
  There is no standardized definition of prolonged air leak but the investigators' previous analyses have focused on 48 hours as a cut-off. Around 50% of adolescents treated for primary spontaneous pneumothorax suffer from this complication leading to prolonged hospital stays and increased hospital costs, as well as impacting patient mental health.
Procedural Pain score | 30 days
  Due to concerns that the algorithm may impact patient pain, the investigators will gather data on postoperative pain scores used by nursing staff to evaluate need for additional pain medication. Nursing staff use a Numerical Rating Scale where the minimum value is 1 and the maximum value is 10, with 10 being the worst pain.

OTHER OUTCOMES:
Incidence of Infectious Complications | 30 days
  Although not seen in the pediatric literature, adult literature has described a case of empyema after autologous blood patch. The investigators will therefore keep track of any of these negative outcomes in this pilot study.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Gulack, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No